CLINICAL TRIAL: NCT00614653
Title: Phase I Trial of Preoperative Radiotherapy With Concurrent Bevacizumab, Erlotinib and Capecitabine for Locally Advanced Pancreatic Cancer
Brief Title: Bevacizumab, Erlotinib and Capecitabine for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0044; NCI-2010-01549 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Bevacizumab; Avastin™; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Erlotinib; Erlotinib Hydrochloride; Tarceva; OSI-774; Capecitabine; Xeloda
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab, Erlotinib + Capecitabine (Experimental): Bevacizumab intravenous (IV) every 2 weeks at 5 mg/kg, Erlotinib 100 mg orally (PO) daily + Capecitabine 400 mg/m2 PO twice daily (BID) only on days of radiation. Radiation treatment once daily for 5 1/2 weeks or 28 doses, Dose 50.4 Gy.
  Interventions: Drug: Bevacizumab; Drug: Erlotinib; Drug: Capecitabine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg IV Over 90 Minutes Every 2 Weeks
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Erlotinib — 100 mg by mouth Once Daily on days with radiation.
  Other Names: OSI-774; Tarceva
Drug: Capecitabine — 400 mg/m^2 PO Twice Daily on days with radiation.
  Other Names: Xeloda
Radiation: Radiation Therapy — Radiation treatment once daily for 5 1/2 weeks or 28 doses, Dose 50.4 Gy
  Other Names: XRT; RT; radiotherapy

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of capecitabine, erlotinib hydrochloride, and bevacizumab that can be given in combination with radiation to patients with pancreatic cancer.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

Capecitabine and erlotinib hydrochloride are designed to interfere with the growth of cancer cells.

Study Drug Dose Level:

If you are found to be eligible to take part in the study, you will begin receiving capecitabine, erlotinib hydrochloride, and bevacizumab. The dose you receive will be based on how many participants have been enrolled before you, and on the safety data that are available. The first group of enrolled participants will be given low doses of capecitabine, erlotinib hydrochloride, and bevacizumab. If no intolerable side effects occur, the next group will be enrolled at a higher dose level. This process will continue until researchers find the highest dose of capecitabine, erlotinib hydrochloride, and bevacizumab that can be given without intolerable side effects occurring. The study doctor will tell you what dose you will be receiving and how it compares to the doses other participants have received.

Study Drug Administration:

On Days 1, 14, and 28, you will receive bevacizumab through a needle in your vein. Your first infusion will last about 90 minutes. If you tolerate the drug well, the next infusion will last about 60 minutes. If the 60-minute infusion is well tolerated, all other infusions will last about 30 minutes.

On each day that you receive radiation, you will take capecitabine and erlotinib hydrochloride by mouth in the morning and evening with food.

Radiation:

You will receive radiation once a day on Monday through Friday, excluding holidays. This schedule will be continue for 5 1/2 weeks or 28 doses.

Study Visits:

Every week while you are on study, you will have the following tests and procedures performed:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked about any side effects you may be experiencing.
* You will repeat the same health questionnaire that you filled out at screening.

Bevacizumab and Surgery:

If at any time during the study the tumor can be removed surgically, you will have surgery. A separate consent form would be used. Because bevacizumab may slow the healing of wounds, study participants may not have surgery within 10 weeks after the last bevacizumab infusion.

Length of Study:

You will remain on study for up to 5 1/2 weeks. You will be taken off-study early if the disease gets worse or intolerable side effects occur.

End-Of-Study Visit:

Four (4) to 6 weeks after you finish radiation, you will have an end-of-study visit with the following tests and procedures performed:

* You will have a complete physical exam.
* Blood (about 2 tablespoons) and urine will be collected for routine tests.
* You will have chest x-rays and CT scans of the abdomen.
* You will repeat the health questionnaire.

Additional Experimental Therapy:

If you appear to be benefitting from the experimental therapy, the study doctor may decide to continue your experimental therapy after the end-of-study visit. This would be daily erlotinib hydrochloride, with bevacizumab infusions every 2 weeks unless the disease gets worse or intolerable side effects occur. You would have study visits once a month, with the same procedures as you did during the weekly study visits (except for the questionnaires).

This is an investigational study. Capecitabine, bevacizumab, and erlotinib hydrochloride are FDA approved and commercially available. The use of capecitabine and bevacizumab for pancreatic cancer and in combination with erlotinib hydrochloride is investigational. At this time, the 3-drug combination is being used in research only.

Up to 30 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status of 0 or 1.
2. Patients must be >/= 18 years of age. There will be no upper age restriction.
3. Cytologic or histologic proof of adenocarcinoma of the pancreas. Patients can have tumor originating in any part of the pancreas. Islet cell tumors are not eligible. Only patients with non- metastatic, unresectable disease are eligible. Patients who cannot undergo resection because of underlying medical problems are also eligible. Patients with regional nodal disease are eligible.
4. All patients must be staged with a physical exam, CXR, and contrast-enhanced helical thin-cut abdominal CT. Unresectability is defined by CT criteria: a) evidence of tumor extension to the celiac axis or superior mesenteric (SM) artery, or b) evidence on either CT or angiogram of occlusion of the SM vein or SM/ portal vein confluence. If a tumor does not meet this definition and is found to be unresectable at surgical exploration, then that tumor is considered unresectable.
5. Patients may have received prior chemotherapy but not prior radiation therapy to the upper abdomen.
6. Bone marrow function: absolute neutrophil count (ANC) >1,500/ul. Platelets >100,000/ul.
7. Hepatic function: Total bilirubin less than 5mg/dL. If the patient required an endobiliary stent, the bilirubin level must have declined on consecutive measurements indicating adequate biliary decompression; alanine aminotransferase (ALT) </= 5 times the upper limit of normal.
8. Renal function: BUN </= 30 mg%, creatinine </= 1.5 mg% and creatinine clearance >/= 30ml/min (estimated as calculated with Cockcroft-Gault equation). Note: In patients with moderate renal impairment (estimated creatinine clearance 30-50 mL/min) at baseline, a dose reduction to 75% of the capecitabine starting dose is recommended.
9. Patients must have signed informed consent indicating that they are aware of the investigational nature of the study, and are aware that participation is voluntary.

Exclusion Criteria:

1. Prior abdominal radiotherapy.
2. Imaging (CT or MRI) or endoscopic evidence of direct duodenal invasion by tumor.
3. Prior therapy with bevacizumab, cetuximab, or gefitinib. Prior therapy with erlotinib is permitted unless the patient was taken off erlotinib due to treatment failure.
4. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in any other experimental drug study.
5. Prior severe infusion reaction (bronchospasm, stridor, urticaria and/or hypotension) to a monoclonal antibody.
6. Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil.
7. Proteinuria at baseline or clinically significant impairment of renal function as demonstrated by urine dipstick for proteinuria >/= 2+ (patients discovered to have >/= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible).
8. Prior history of cancer within the last five years except for basal cell carcinoma of the skin or carcinoma in situ of the cervix. Patients with previous malignancies but without evidence of disease for 5 years will be allowed to enter the trial.
9. Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Women / men of childbearing potential not using a reliable contraceptive method (oral contraceptive , other hormonal contraceptive, intrauterine device, diaphragm or condom). (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients must agree to continue contraception for 30 days from the date of the last study drug administration.
10. Serious, uncontrolled, concurrent infection(s) requiring IV antibiotics or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy.
11. Uncontrolled hypertension [blood pressure of >/=140/90 mmHg on medication], New York Heart Association (NYHA) Class II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), significant vascular disease (e.g., aortic aneurysm, aortic dissection) or Class II or greater peripheral vascular disease, history of stroke or TIA within 6 months prior to study enrollment, history of hypertensive crisis or hypertensive encephalopathy.
12. History of active angina or myocardial infarction within 6 months. History of significant ventricular arrhythmia requiring medication with antiarrhythmics, or a history of a clinically significant conduction system abnormality.
13. Psychiatric disorders rendering patients incapable of complying with the requirements of the protocol.
14. History or evidence upon physical examination of CNS disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of stroke)
15. Prior history of pulmonary embolism or deep venous thrombosis.
16. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study, other than that defined by protocol; fine needle aspirations or core biopsies within 7 days prior to Day 0.
17. Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome or inability to swallow.
18. Known, existing uncontrolled coagulopathy, INR >/= 1.5.
19. Patients on Coumadin must be changed to Lovenox at least 1 week prior to starting capecitabine. Low dose (1 mg) Coumadin is allowed. Intravenous and low-molecular weight heparin are permitted.
20. Patients taking Sorivudine or Brivudine must be off of these drugs for 4 weeks prior to starting capecitabine. Patients taking cimetidine must have this drug discontinued. Ranitidine or a drug from another anti-ulcer class can be substituted for cimetidine if necessary. If patient is currently receiving allopurinol, must discuss with PI to see of another agent may substitute for it.
21. Current serious, nonhealing wound, ulcer, or bone fracture.
22. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0.
23. Patients who have had an organ allograft.
24. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Highest Tolerated Dose of Capecitabine, Erlotinib Hydrochloride, and Bevacizumab + Radiation | 5 1/2 Weeks
  Any of these events considered a dose-limiting toxicity.
  1. Any grade 4 hemorrhage, grade 2 pulmonary or CNS hemorrhage
  2. Cardiac arrhythmia
  3. Grade 4 congestive heart failure
  4. Grade 4 hypertension or reversible posterior leukoencephalopathy syndrome (RPLS)
  5. Grade 4 nephrotic syndrome
  6. Grade 4 diarrhea
  7. Grade 4 rash
  8. Pulmonary adverse event related to erlotinib
  9. Bowel perforation
  10. Symptomatic Grade 4 venous thromboembolic event, or any grade arterial thromboembolic event
  11. Wound dehiscence requiring medical or surgical intervention
  12. Determination by the investigator that it is no longer safe for the subject to continue therapy

SECONDARY OUTCOMES:
Response Rate of Addition of Bevacizumab and Erlotinib to Capecitabine-Based Chemoradiation | 4 to 6 weeks after radiation treatment
  Complete response (CR) - complete disappearance of clinical evidence of a tumor. Partial response (PR) - 50% or greater decrease in sum of products of the longest perpendicular diameters of all measured lesions compared to baseline. Stable disease (SD) - no significant change in disease status. Progressive disease (PD) - a 25% increase in the area of malignant lesions >2 cm2 or in sum of products of the longest perpendicular diameters of individual lesions in a given organ site. If only one lesion is available for measurement, a 50% increase in the size if the area of the lesion was 2 cm2. The appearance of new lesions will also constitute progressive disease. Comparisons of tumor size made with previous smallest measurement in patients who have attained a partial response or with baseline measurements in patients with stable disease. Tumor progression also defined as significant clinical deterioration that cannot be attributed to treatment or other medical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Krishnan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org